CLINICAL TRIAL: NCT03409107
Title: A 28-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center, Study in Recombinant Human Erythropoietin (rhEPO) naïve Non-dialysis Participants With Anemia Associated With Chronic Kidney Disease to Evaluate the Efficacy, Safety and Effects on Quality of Life of Daprodustat Compared to Placebo
Brief Title: Anemia Studies in Chronic Kidney Disease (CKD): Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor (PHI) Daprodustat in Non-Dialysis Subjects Evaluating Hemoglobin (Hgb) and Quality of Life (ASCEND-NHQ)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205270; 2017-002270-39 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Anaemia
Keywords: Non-Dialysis; Anemia; Chronic kidney disease; Recombinant human erythropoietin naïve; Hemoglobin; Daprodustat
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive Daprodustat or placebo in a randomized manner.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. The participant, investigator, site staff, and study team will be blinded to the assigned study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daprodustat receivers (Experimental): Participants will receive oral daprodustat once daily
  Interventions: Drug: Daprodustat (GSK1278863); Drug: Iron therapy
- Placebo receivers (Placebo Comparator): Participants will receive oral placebo once daily
  Interventions: Drug: Placebo; Drug: Iron therapy

INTERVENTIONS:
Drug: Daprodustat (GSK1278863) — Daprodustat will be available as 9 millimeter (mm) or 7 mm film-coated tablets. Daprodustat will be administered once daily via oral route and can be taken without regard to food.
  Arms: Daprodustat receivers
Drug: Placebo — Daprodustat matching placebo will be available as 9 mm or 7 mm film coated tablets. Placebo will be administered once daily via oral route and can be taken without regard to food.
  Arms: Placebo receivers
Drug: Iron therapy — Iron therapy will be administered if ferritin is <50 Nano gram per milliliter and/or TSAT is <15 percent.

SUMMARY:
The purpose of this multi-center study in non-dialysis participants with anemia associated with CKD is to evaluate safety, efficacy and quality of life of daprodustat compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age at the time of signing the informed consent.
* Have CKD, confirmed at screening: Kidney Disease Outcomes Quality Initiative (KDOQI) CKD stages 3, 4, or 5 defined by Estimated glomerular filtration rate (eGFR) using the CKD Epidemiology Collaboration (CKD-EPI) formula.
* Participants with Stable HemoCue Hgb from 8.5 to 10.5 at screening visit (Week -4) and from 8.5 to 10.0 g/dL at randomization (Day 1).
* Participants may receive up to one intravenous (IV) iron dose within the 8 weeks prior to screening and NO IV iron use between screening visit and randomization (Day 1).
* If needed, participant may be on stable maintenance oral iron supplementation. There should be <50% change in overall dose and no change in type of iron prescribed in the 4 weeks prior to Day 1 randomization visit.
* Male and female participants are eligible. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 weeks after the last dose of study treatment.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participants who are on dialysis or clinical evidence of impending need to initiate dialysis within 180 days after randomization (Day 1).
* Planned living-related or living-unrelated kidney transplant within 28 weeks after randomization (Day 1).
* Transferrin saturation (TSAT) <15 percent (Screening only).
* Ferritin <50 nanograms per milliliter (ng/mL) (Screening only).
* History of rhEPO or rhEPO analogue use within the 8 weeks prior to screening and rhEPO use between screening and randomization (Day 1).
* History of transfusion within the 8 weeks prior to screening and transfusion between screening and randomization (Day 1).
* History of bone marrow aplasia or pure red cell aplasia (PRCA).
* Participants with Megaloblastic anemia (untreated pernicious anemia and folate deficiency), thalassemia major, sickle cell disease or myelodysplastic syndrome.
* Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant gastrointestinal (GI) bleeding <= 8 weeks prior to screening through to randomization (Day 1).
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
* Use of strong inhibitor of CYP2C8 (for example, gemfibrozil) or strong inducers of CYP2C8 (for example, rifampin/rifampicin).
* Ferric citrate use within 4 weeks prior to randomization (Day 1).
* Use of other investigational agent or device prior to screening through to randomization (Day 1).
* Any prior treatment with daprodustat for a treatment duration of >30 days.
* MI or acute coronary syndrome within the 8 weeks prior to screening through to randomization. (Day 1).
* Stroke or transient ischemic attack within the 8 weeks prior to screening through to randomization. (Day 1).
* Chronic Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* QT interval corrected by Bazett's formula (QTcB) >500 milliseconds (msec) or QTcB >530 msec in participants with bundle branch block. There is no corrected QT interval (QTc) exclusion for participants with a predominantly paced rhythm.
* Alanine transaminase (ALT) >2x upper limit of normal (ULN) at screening (Week -4).
* Bilirubin >1.5xULN at screening (Week -4).
* Current unstable liver or biliary disease per investigator assessment, generally defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* History of malignancy within the 2 years prior to screening through to randomization (Day 1), or currently receiving treatment for cancer, or complex kidney cyst (for example, Bosniak Category II F, III or IV) > 3 centimeters (cm).
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the participant at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.
* Current uncontrolled hypertension as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (148):
- United States (47):
  - GSK Investigational Site, Homewood, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Downey, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Lynwood, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Salinas, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Statesboro, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Buckley, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Brookhaven, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Rochester, New Hampshire
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Midwest City, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Scottdale, Pennsylvania
  - GSK Investigational Site, Smithfield, Pennsylvania
  - GSK Investigational Site, West Reading, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, DeSoto, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Waxahachie, Texas
  - GSK Investigational Site, Norfolk, Virginia
- Argentina (6):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Nicolás de los Arroyos, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe
- Australia (5):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Fitzroy
- Brazil (8):
  - GSK Investigational Site, Vitória, Espírito Santo
  - GSK Investigational Site, Feira de Santana, Estado de Bahia
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, Santo André - SP, São Paulo
  - GSK Investigational Site, São Bernardo do Campo, São Paulo
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, São Paulo
- Canada (11):
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- France (8):
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Melun
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Saint-Priest-en-Jarez
- Italy (7):
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Mestre, Veneto
- Mexico (9):
  - GSK Investigational Site, León, Guanajuato
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Boca del Rio, Veracruz
  - GSK Investigational Site, Córdoba, Veracruz
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Veracruz
- Poland (12):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Ciechanów
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Oława
  - GSK Investigational Site, Pleszew
  - GSK Investigational Site, Sosnowiec
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Świdnik
  - GSK Investigational Site, Tczew
  - GSK Investigational Site, Warsaw
- Romania (8):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Târgu Mureş
  - GSK Investigational Site, Timișoara
- Russia (12):
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kaliningrad
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Yaroslavl
- South Korea (5):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (7):
  - GSK Investigational Site, Canterbury, Kent
  - GSK Investigational Site, Derby
  - GSK Investigational Site, London
  - GSK Investigational Site, Peterborough
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Shrewsbury
  - GSK Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Johansen KL, Cobitz AR, Singh AK, Macdougall IC, Lopes RD, Obrador GT, Kovesdy CP, Israni R, Jha V, Okoro T, Sprys M, Jolly S, Lindsay AC, Bhatt P, Camejo RR, Keeley T, Cizman B, Wheeler DC. The ASCEND-NHQ randomized trial found positive effects of daprodustat on hemoglobin and quality of life in patients with non-dialysis chronic kidney disease. Kidney Int. 2023 Jun;103(6):1180-1192. doi: 10.1016/j.kint.2023.02.019. Epub 2023 Mar 2. PMID 36868377
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 142 centers in 14 countries. Participants were randomized to receive either Daprodustat or Placebo.
Pre-assignment Details: A total of 1336 participants were screened, of which 722 were screen failures. A total of 614 participants were enrolled in the study.
Groups:
- Placebo: Participants received matching placebo once daily orally for up to 28 weeks followed by 4 weeks of follow-up.
- Daprodustat: Participants received daprodustat tablets with titrated dose levels ranging from 1, 2, 4, 6, 8, 10, 12, 16 milligrams (mg) once daily orally for up to 28 weeks, followed by 4 weeks of follow-up. Study treatment was dose-titrated to achieve and maintain hemoglobin in the target range (11 to 12 grams per deciliter [g/dL])
Period: Overall Study
Arm/Group | Placebo | Daprodustat
Started | 307 | 307
Completed | 290 | 300
Not Completed | 17 | 7
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 7 | 2
Not completed — Adverse Event | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Daprodustat | Total
Number analyzed (Participants) | 307 | 307 | 614
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (12.93) | 65.3 (13.43) | 65.9 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 176 | 354
  Male | 129 | 131 | 260
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 34 | 34 | 68
  ASIAN: CENTRAL/SOUTH ASIAN HERITAGE | 3 | 6 | 9
  ASIAN: JAPANESE/EASTASIAN/SOUTHEAST ASIAN HERITAGE | 24 | 24 | 48
  ASIAN: MIXED ASIAN RACE | 1 | 0 | 1
  BLACK OR AFRICAN AMERICAN | 47 | 44 | 91
  NATIVE HAWAIIAN/OTHER PACIFIC ISLANDER | 1 | 0 | 1
  WHITE | 195 | 197 | 392
  BLACK OR AFRICAN AMERICAN AND WHITE | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin From Baseline and Over the Evaluation Period (Mean Over Week 24 and 28)
Description: Blood samples were collected at given time points from participants for hemoglobin measurements. Evaluation period hemoglobin value was defined as the mean of all available post-randomization hemoglobin values (on and off-treatment) during the evaluation period (Week 24 to Week 28 inclusive). For the primary analysis, the missing post-Baseline hemoglobin values were imputed using pre-specified multiple imputations. Change from Baseline was defined as the average of post-randomization values during the evaluation period minus Baseline value. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using the Analysis of Covariance (ANCOVA) model with terms for treatment, Baseline hemoglobin, and region.
Time Frame: Baseline (Day 1) and Week 24 to Week 28
Population: Intent-to-Treat (ITT) Population comprised all randomized participants regardless of whether they took study drug.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 307 | 307
Grams per deciliter | 0.19 (0.062) | 1.58 (0.061)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p < 0.0001, ANCOVA; One-sided p-value based on test of null hypothesis: (Daprodustat - Placebo) <= 0 versus alternative: difference > 0; LS Mean Difference = 1.40, 95% CI 2-sided [1.23 to 1.56] — Treatment group comparisons were based on a ANCOVA model with terms for treatment, Baseline hemoglobin, and region

2. Secondary Outcome: Percentage of Participants With Hemoglobin Increase of >=1.0 Grams Per Deciliter From Baseline to Evaluation Period
Description: Blood samples were collected at given time points for hemoglobin measurements. Evaluation period hemoglobin value was defined as the mean of all available post-randomization hemoglobin values (on and off-treatment) during the evaluation period (Week 24 to Week 28 inclusive). For the primary analysis, the missing post-Baseline hemoglobin values were imputed using pre-specified multiple imputations. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date. Percentage of participants with hemoglobin increase of >=1.0 grams per deciliter from Baseline to evaluation period was analyzed using Cochran-Mantel-Haenszel (CMH) chi-squared test. The percentage values presented has been rounded off.
Time Frame: Baseline (Day 1) and Week 24 to Week 28
Population: Intent-to-Treat population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 307 | 307
Percentage of participants | 18 | 77
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — One-sided p-value was based on test of null hypothesis: (Daprodustat - Placebo) <=0 versus alternative: difference > 0; Difference in Response rate = 0.56, 95% CI 2-sided [0.49 to 0.63] — Treatment group comparisons were based on a Cochran-Mantel-Haenszel test adjusted for treatment group and region

3. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Questionnaire Vitality Domain Score by Traditional Scoring at Week 28
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the 8 health domains: Physical Functioning, Role-Physical (role limitations caused by physical problems), Social Functioning, Bodily Pain, Mental Health, Role-Emotional (role limitations caused by emotional problems), Vitality, and General Perception of Health.Each domain is scored from 0 (poorer health) to 100 (better health). Vitality domain score ranges from 0-100; higher score indicates a better health state & better functioning. Change from Baseline was calculated as Post-Dose Visit Value at Week 28 minus Baseline. For primary analysis, the missing on-treatment Week 28 SF-36 Vitality domain scores were imputed using pre-specified multiple imputations. Baseline value was latest non-missing pre-dose assessment on or before randomization date. Analysis was performed using ANCOVA model with terms for treatment, Baseline score, and region.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 307 | 307
Scores on a scale | 1.93 (1.161) | 7.29 (1.121)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0005, ANCOVA — One-sided p-value based on test of null hypothesis:(Daprodustat-Placebo) <= 0 vs alternative: difference > 0; LS Mean Difference = 5.36, 95% CI 2-sided [2.17 to 8.56] — Treatment group comparisons were based on ANCOVA model with terms for treatment, Baseline score, and region

4. Secondary Outcome: Percentage of Participants With Hgb Response (Hgb in the 11-12 Grams/Deciliter Range) During Evaluation Period (Week 24 to Week 28 Inclusive)
Description: Mean hemoglobin during the evaluation period was defined as the mean of all evaluable hemoglobin values during the evaluation period (Week 24 to Week 28 inclusive) including any evaluable unscheduled hemoglobin values that were taken during this period. Percentage of participants with Hgb response was defined as participants with mean Hgb within range (11-12 grams per deciliter during the evaluation period (Week 24 to Week 28 inclusive) and it was analyzed using Cochran-Mantel-Haenszel (CMH) chi-squared test. The percentage values presented has been rounded off.
Time Frame: Week 24 to Week 28
Population: Intent-to-Treat Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 307 | 307
Percentage of participants | 8 | 52
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Difference in Response rate = 0.45, 95% CI 2-sided [0.37 to 0.52] — Treatment group comparisons are based on a Cochran-Mantel-Haenszel test adjusted for treatment group, and region

5. Secondary Outcome: Percentage of Time With Hgb Within the Target Range (11-12 Grams Per Deciliter) During Evaluation Period (Week 24 to Week 28 Inclusive) (Hodges-Lehmann Estimate)
Description: Percentage of days for which participant's Hgb was within the target range of 11-12 grams per deciliter during the evaluation period (Week 24 to Week 28 inclusive), including any unscheduled evaluable Hgb values that were taken during this time period. Percentage of time for which Hgb was within the target range (11-12 grams per deciliter) for a participant was calculated by dividing 'the total number of days that Hgb was within range during Week 24 to 28' by 'the total number of days the participant remained on treatment during Week 24 to 28'.
Time Frame: Week 24 to Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 216 | 252
Percentage of days | 0.00 [0.0 to 100.0] | 53.59 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; Hodges-Lehmann Estimate; Hodges-Lehmann Estimate of treatment difference has been reported; Difference in treatment effect = 38.80, 95% CI 2-sided [25.00 to 54.55]

6. Secondary Outcome: Percentage of Time With Hgb Within the Target Range (11-12 Grams Per Deciliter) During Evaluation Period (Week 24 to Week 28 Inclusive) (Mann-Whitney Estimate)
Description: as for outcome 5
Time Frame: Week 24 to Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 216 | 252
Percentage of days | 0.00 [0.0 to 100.0] | 53.59 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p < 0.0001, van Elteren test — One-sided superiority p-value from the van Elteren test; Difference in treatment effect = 0.768, 95% CI 2-sided [0.729 to 0.806] — Mann-Whitney estimate of the treatment difference stratified by region has been presented

7. Secondary Outcome: Change From Baseline in Post-randomization Hgb at Week 28
Description: Blood samples were collected at given time points for hemoglobin measurements. Change from Baseline in Hgb was analyzed using a mixed model repeated measures (MMRM) approach. Change from Baseline was calculated as Post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 301 | 299
Grams per deciliter | 0.20 (0.070) | 1.56 (0.069)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p < 0.0001, MMRM — One-sided superiority p-value from the MMRM model; LS Mean difference = 1.36, 95% CI 2-sided [1.16 to 1.55] — Treatment group comparisons were based on MMRM fitted from Baseline up to Week 28, with factors for treatment, time, region, Baseline Hb and Baseline Hb by time and treatment by time interactions

8. Secondary Outcome: Rate of Participants Permanently Stopping Randomized Treatment Due to Meeting Rescue Criteria
Description: The incidence rate of participants permanently stopping randomized treatment due to meeting rescue criteria is presented.
Time Frame: Up to Week 28
Population: Intent-to-Treat Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person year
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 307 | 307
Events per 100 person year | 18.88 [12.33 to 27.66] | 1.33 [0.16 to 4.82]
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0002, Wald test — One-sided p-value was based on Wald test of null hypothesis: (Daprodustat/Placebo) >=1 versus alternative: ratio<1; Hazard Ratio (HR) = 0.07, 95% CI 2-sided [0.02 to 0.30] — Hazard ratio was estimated using a Cox proportional hazard regression model adjusted for treatment group and region

9. Secondary Outcome: Change From Baseline by Domain and Single Item Scores on the Chronic Kidney Disease -Anemia Questionnaire (CKD-AQ) Symptom Questionnaire
Description: CKD-AQ is 21-item patient reported outcomes measure assessing symptoms & symptom impact in participants with anemia associated with CKD.CKD-AQ identified 3 domains:1.Tired/Low Energy/Weak scale consisting of ten items;2.Chest Pain/Shortness of Breath scale consisting of four items and 3.Cognitive scale consisting of three items;Single items included: 4.Difficulty Sleeping;5.Difficulty Standing for long periods of time;6.Severity-Shortness of breath while sitting/resting;7.Time with Shortness of breath while not doing activity.Single-item measures were recorded based on 0-100 scoring with 0 is worst possible & 100 is best possible score.Total domain score is calculated as average of items in each domain & ranged from 0-100 where 0 is worst possible and 100 is best possible score.Change from Baseline was calculated as post-dose visit value minus Baseline.Baseline was latest non-missing pre-dose assessment on or before randomization date. Adjusted mean & standard error is presented.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 193 | 212
Scores on a scale
  Tired/Low Energy/Weak Domain | 2.81 (1.132) | 8.72 (1.086)
  Chest Pain/Shortness of Breath Domain | 0.62 (0.971) | 3.55 (0.932)
  Cognitive Domain | 0.48 (1.042) | 4.27 (0.999)
  Difficulty in Sleeping | 2.61 (1.643) | 5.22 (1.577)
  Difficulty Standing for Long Periods of Time | 1.55 (1.630) | 6.19 (1.563)
  Severity-Shortness of Breath, Sitting/Resting | 0.43 (0.995) | 3.11 (0.954)
  Time with Shortness of BreathnotDoingActivity | 0.29 (1.083) | 2.30 (1.037)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p < 0.0001, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 5.91, 95% CI 2-sided [2.83 to 9.00] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Tired/Low Energy/Weak domain
Statistical Analysis 2: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0152, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 2.93, 95% CI 2-sided [0.28 to 5.57] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Chest Pain/Shortness of Breath Domain
Statistical Analysis 3: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0045, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 3.79, 95% CI 2-sided [0.95 to 6.63] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Cognitive Domain
Statistical Analysis 4: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.1267, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 2.61, 95% CI 2-sided [-1.87 to 7.09] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Difficulty Sleeping
Statistical Analysis 5: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0203, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 4.64, 95% CI 2-sided [0.20 to 9.09] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Difficulty Standing for Long Periods of Time
Statistical Analysis 6: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0266, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 2.68, 95% CI 2-sided [-0.04 to 5.39] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Severity of Shortness of Breath While Sitting or Resting
Statistical Analysis 7: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0907, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 2.01, 95% CI 2-sided [-0.94 to 4.96] — Analysis was performed by MMRM with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Time with Shortness of Breath While not Doing an Activity

10. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S)
Description: The PGI-S is a 1-item questionnaire designed to assess participant's impression of disease severity on a 5-point disease severity scale (0=absent, 1=mild, 2=moderate, 3=severe, or 4=very severe). A higher score indicated worse outcome. Change from Baseline was calculated as Post-Dose visit value minus Baseline value. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 193 | 212
Scores on a scale | -0.04 (0.055) | -0.18 (0.052)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0391, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-rhEPO) >=0 versus alternative: difference <0; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.28 to 0.02] — MMRM fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions

11. Secondary Outcome: Change From Baseline in the SF-36 Physical Functioning Domain
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following eight health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality, and general perception of health. Each domain is scored from 0 (poorer health) to 100 (better health). Physical functioning domain score ranges from 0-100; higher score indicates a better health state and better functioning. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 190 | 210
Scores on a scale | 1.23 (1.354) | 3.80 (1.298)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0858, MMRM — One sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 vs. alternative: difference >0; Mean Difference (Net) = 2.57, 95% CI 2-sided [-1.12 to 6.26] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Change From Baseline of the SF-36 Individual Items in the Vitality Domain
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following eight health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality, and general perception of health. Individual vitality items include: 1. Did you feel full of life?, 2. Did you have a lot of energy?, 3. Did you feel worn out?, 4. Did you feel tired?. Score of each item in the vitality domain ranges from 0-100; higher score indicates better health state and better functioning. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 190 | 210
Scores on a scale
  Did you feel full of life? | -0.02 (0.070) | 0.16 (0.067)
  Did you have a lot of energy? | 0.09 (0.066) | 0.26 (0.063)
  Did you feel worn out? | 0.16 (0.067) | 0.34 (0.064)
  Did you feel tired? | 0.08 (0.060) | 0.34 (0.057)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0357, MMRM — One sided p-value based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.02 to 0.36] — MMRM fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Did you feel full of life?
Statistical Analysis 2: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0328, MMRM — One-sided p-value based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.01 to 0.35] — MMRM fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Did you have a lot of energy?
Statistical Analysis 3: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0252, MMRM — One-sided p-value based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 0.18, 95% CI 2-sided [0.00 to 0.37] — MMRM fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Did you feel worn out?
Statistical Analysis 4: Comparison: Placebo; Test type: Superiority; p = 0.0010, MMRM — One-sided p-value based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus alternative: difference >0; Mean Difference (Net) = 0.26, 95% CI 2-sided [0.10 to 0.42] — MMRM fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions for Did you feel tired?

13. Secondary Outcome: Number of Participants Currently Employed as Per Work Productivity and Activity Impairment Questionnaire: Anemic Symptoms Clinical Practice Version (WPAI-ANS-CPV)
Description: WPAI-ANS-CPV is anemia specific questionnaire designed as self-reported quantitative assessment of social functioning related to work and regular daily activities. It contains 2 concepts-work productivity impairment measured via absenteeism(time missed from work), presenteeism(impairment at work) and regular daily activity impairment. WPAI questions (Q) were:1) currently employed,2) work time missed due to problem, 3) impairment while working due to problem, 4) overall work impairment due to problem, 5) activity impairment due to problem. WPAI generates 4 domain scores:percent (%) of work time missed(absenteeism),% of impairment while working(presenteeism),% of overall work impairment(absenteeism and presenteeism combined),% of activity impairment. Number of participants currently employed as per WPAI-ANS-CPV is presented.
Time Frame: Week 8, Week 12 and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 249 | 251
Participants
  Week 8, No, n=249, 250: number analyzed (Participants) | 249 | 250
  Week 8, No, n=249, 250 | 195 | 204
  Week 8, Yes, n=249, 250: number analyzed (Participants) | 249 | 250
  Week 8, Yes, n=249, 250 | 54 | 46
  Week 12, No, n=234, 251: number analyzed (Participants) | 234 | 251
  Week 12, No, n=234, 251 | 183 | 212
  Week 12, Yes, n=234, 251: number analyzed (Participants) | 234 | 251
  Week 12, Yes, n=234, 251 | 51 | 39
  Week 28, No, n=193, 213: number analyzed (Participants) | 193 | 213
  Week 28, No, n=193, 213 | 158 | 178
  Week 28, Yes, n=193, 213: number analyzed (Participants) | 193 | 213
  Week 28, Yes, n=193, 213 | 35 | 35

14. Secondary Outcome: Change From Baseline in WPAI-ANS-CPV: Percent Time Missed From Work
Description: WPAI-ANS-CPV is anemia specific questionnaire designed as self-reported quantitative assessment of social functioning related to work and regular daily activities. It contains 2 concepts-work productivity impairment measured via absenteeism (time missed from work), presenteeism (impairment at work) and regular daily activity impairment. WPAI questions (Q) were: 1) currently employed, 2) work time missed due to problem, 3) impairment while working due to problem, 4)overall work impairment due to problem, 5) activity impairment due to problem. Percent work time missed due to problem was a subscale and calculated as: Q2/(Q2+Q4) for those who were currently employed. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment and less productivity. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Week 8, Week 12 and Week 28
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 50 | 39
Percentage of time
  Week 8, n=50, 39 | -2.4 (28.40) | -6.1 (24.92)
  Week 12, n=46, 31: number analyzed (Participants) | 46 | 31
  Week 12, n=46, 31 | 0.9 (28.79) | 4.2 (27.96)
  Week 28, n=28, 25: number analyzed (Participants) | 28 | 25
  Week 28, n=28, 25 | 0.0 (33.59) | 0.3 (31.01)

15. Secondary Outcome: Change From Baseline in WPAI-ANS-CPV: Mean Hours Missed From Work in the Past 7 Days
Description: WPAI-ANS-CPV is anemia specific questionnaire designed as self-reported quantitative assessment of social functioning related to work and regular daily activities. It contains 2 concepts-work productivity impairment measured via absenteeism (time missed from work), presenteeism (impairment at work) and regular daily activity impairment. WPAI Qs were: 1) currently employed, 2) work time missed due to problem, 3) impairment while working due to problem, 4) overall work impairment due to problem, 5) activity impairment due to problem. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Week 8, Week 12 and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at indicated time points are presented (presented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Percentage of hours
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 50 | 39
Percentage of hours
  Week 8, n=50, 39 | 0.1 (18.46) | -1.8 (11.88)
  Week 12, n=46, 31: number analyzed (Participants) | 46 | 31
  Week 12, n=46, 31 | 1.4 (14.07) | 2.4 (16.83)
  Week 28, n=28, 25: number analyzed (Participants) | 28 | 25
  Week 28, n=28, 25 | 0.3 (19.90) | 1.0 (14.24)

16. Secondary Outcome: Change From Baseline in WPAI: Percent Impairment at Work
Description: WPAI-ANS-CPV is anemia specific questionnaire designed as self-reported quantitative assessment of social functioning related to work and regular daily activities.It contains 2 concepts-work productivity impairment measured via absenteeism(time missed from work),presenteeism(impairment at work) and regular daily activity impairment.WPAI Qs were:1)currently employed,2)work time missed due to problem,3)impairment while working due to problem,4)overall work impairment due to problem,5)activity impairment due to problem. % Impairment while Working due to Problem was subscale and calculated as: Q5/10 for those who were currently employed and actually worked in past 7 days. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment and less productivity. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before randomization date.
Time Frame: Baseline (Day 1), Week 8, Week 12 and Week 28
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 45 | 32
Percentage of impairment
  Week 8, n=45, 32 | -5.1 (18.42) | -11.3 (24.06)
  Week 12, n=41, 26: number analyzed (Participants) | 41 | 26
  Week 12, n=41, 26 | -4.6 (18.99) | -8.8 (23.38)
  Week 28, n=24, 20: number analyzed (Participants) | 24 | 20
  Week 28, n=24, 20 | -9.6 (25.62) | -9.0 (22.92)

17. Secondary Outcome: Change From Baseline in WPAI: Percent Overall Work Impairment
Description: WPAI-ANS-CPV is anemia specific questionnaire designed as self-reported quantitative assessment of social functioning related to work and regular daily activities. It contains 2 concepts-work productivity impairment measured via absenteeism (time missed from work), presenteeism (impairment at work) and regular daily activity impairment. WPAI Qs were: 1) currently employed, 2) work time missed due to problem, 3) impairment while working due to problem, 4) overall work impairment due to problem, 5) activity impairment due to problem. Percent overall work impairment due to problem was a subscale and calculated as: Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))×(Q5/10)] for those who were currently employed. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before randomization date.
Time Frame: Baseline (Day 1), Week 8, Week 12 and Week 28
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 45 | 32
Percentage of impairment
  Week 8, n=45, 32 | -4.3 (24.04) | -12.0 (25.90)
  Week 12, n=41, 26: number analyzed (Participants) | 41 | 26
  Week 12, n=41, 26 | 0.5 (25.81) | -3.2 (33.35)
  Week 28, n=24, 20: number analyzed (Participants) | 24 | 20
  Week 28, n=24, 20 | -9.3 (37.45) | -8.4 (19.12)

18. Secondary Outcome: Change From Baseline in WPAI: Percent Regular Daily Activity Impairment
Description: WPAI-ANS-CPV is anemia specific questionnaire designed as self-reported quantitative assessment of social functioning related to work and regular daily activities.It contains 2 concepts-work productivity impairment measured via absenteeism (time missed from work), presenteeism (impairment at work) and regular daily activity impairment. WPAI Qs were: 1) currently employed, 2) work time missed due to problem, 3) impairment while working due to problem, 4) overall work impairment due to problem, 5) activity impairment due to problem. Percent activity impairment due to problem was a subscale and calculated as: Q5/10 for all respondents. Subscale score was expressed as an impairment percentage (range: 0-100%) where higher numbers indicate greater impairment. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before randomization date.
Time Frame: Baseline (Day 1), Week 8, Week 12 and Week 28
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 246 | 248
Percentage of impairment
  Week 8, n=243, 248: number analyzed (Participants) | 243 | 248
  Week 8, n=243, 248 | -4.6 (23.67) | -7.7 (24.53)
  Week 12, n=228, 246: number analyzed (Participants) | 228 | 246
  Week 12, n=228, 246 | -5.2 (25.40) | -8.6 (24.58)
  Week 28, n=187, 210: number analyzed (Participants) | 187 | 210
  Week 28, n=187, 210 | -6.7 (28.93) | -12.2 (27.50)

19. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level Health Utility Index (EQ-5D-5L) Utility Score
Description: The EQ-5D-5L is a self-assessment questionnaire, consisting of 5 items covering 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension is measured by a 5-point Likert scale (1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, and 5: extreme problems). The responses for the five dimension together form a five-figure description of health state. Each of these five-figure health states have attached valuation (utility score), expressed as single index on a scale from 0-1, where 1 is full health and 0 is worst health. The higher the score the better the health status. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at indicated time points are presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 106 | 116
Scores on a scale | 0.01 (0.015) | 0.03 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.1098, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 versus. alternative: difference >0; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.02 to 0.07] — Based on MMRM model fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions

20. Secondary Outcome: Change From Baseline in EuroQol Visual Analogue Scale (EQ-VAS) Score
Description: The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labeled 'the best health you can imagine' and 'the worst health you can imagine' at the time of completion. It is a self-assessment visual analogue scale, ranging from 0=worst imaginable to 100=best. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 106 | 116
Scores on a scale | 0.80 (1.427) | 5.30 (1.373)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0120, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat-Placebo) <=0 vs. alternative: difference >0; Mean Difference (Net) = 4.50, 95% CI 2-sided [0.60 to 8.40] — MMRM model fitted from Baseline up to Week 28 with factors for treatment, time, region, Baseline value and Baseline value by time and treatment by time interactions

21. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Mean Arterial Pressure (MAP) at Week 28
Description: SBP, DBP and MAP were measured with participants in a seated position after at least a 5-minute of rest. MAP is the average BP in an individual's arteries during a single cardiac cycle. Change from Baseline was calculated as post-dose visit value minus Baseline. Baseline value was the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 28
Population: Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 202 | 230
Millimeters of mercury (mmHg)
  SBP | -0.63 (1.045) | -0.23 (0.981)
  DBP | -0.96 (0.625) | 0.84 (0.587)
  MAP | -0.82 (0.674) | 0.49 (0.632)
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.6106, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat - Placebo) >= 0 versus alternative: difference <0; Mean Difference (Net) = 0.40, 95% CI 2-sided [-2.42 to 3.22] — MMRM model fitted from Baseline up to Week 28, with factors for treatment, time, region, Baseline SBP and Baseline SBP by time and treatment by time interactions
Statistical Analysis 2: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.9819, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat - Placebo) >= 0 versus alternative: difference < 0; Mean Difference (Net) = 1.80, 95% CI 2-sided [0.12 to 3.49] — MMRM model fitted from Baseline up to Week 28, with factors for treatment, time, region, Baseline DBP and Baseline DBP by time and treatment by time interactions
Statistical Analysis 3: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.9215, MMRM — One-sided p-value was based on test of null hypothesis: (Daprodustat - Placebo) >= 0 versus alternative: difference <0; Mean Difference (Net) = 1.31, 95% CI 2-sided [-0.51 to 3.13] — MMRM model fitted from Baseline up to Week 28, with factors for treatment, time, region, Baseline MAP and Baseline MAP by time and treatment by time interactions

22. Secondary Outcome: Percentage of Participants With at Least One Blood Pressure (BP) Exacerbation Event
Description: Percentage of participants with at least one BP event is presented. BP exacerbation is defined as: SBP exacerbation: SBP >= 25 mmHg increase from Baseline or SBP >= 180 mmHg; DBP exacerbation: DBP >= 15 mmHg increase from Baseline or DBP >= 110 mmHg. Percentage of participants with at least one BP event is presented. The percentage values presented has been rounded off.
Time Frame: Up to Week 28
Population: Intent-to-Treat Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Daprodustat
Number analyzed (Participants) | 307 | 307
Percentage of participants | 26 | 32
Statistical Analysis 1: Comparison: Placebo vs Daprodustat; Test type: Superiority; p = 0.0680, Cochran-Mantel-Haenszel — One-sided p-value based on test of null hypothesis: (Daprodustat - Placebo) <= 0 versus alternative: difference > 0; Difference in Response rate = 0.06, 95% CI 2-sided [-0.02 to 0.13] — Cochran-Mantel-Haenszel test was performed for treatment group comparison

ADVERSE EVENTS:
Time Frame: All cause mortality, serious adverse events (SAEs) and non-serious AEs were collected up to follow-up (Week 32).
Description: Safety Population comprised of all randomized participants who received at least 1 dose of study treatment. Treatment emergent non-serious adverse events and serious adverse events are reported. One participant who was randomized to placebo accidently received daprodustat during the study and therefore was evaluated in the daprodustat treatment group for the safety outcomes
Arm/Group | Placebo | Daprodustat
All-Cause Mortality (participants affected / at risk) | 16/306 | 10/308
Serious Adverse Events (participants affected / at risk) | 68/306 | 62/308
Other Adverse Events (participants affected / at risk) | 44/306 | 49/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=306) | Daprodustat (N=308)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 5 (6)
Renal failure (Renal and urinary disorders) | 6 (6) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (3) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (4)
Cardiac failure acute (Cardiac disorders) | 4 (4) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 4 (4)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Kidney rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (9) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=306) | Daprodustat (N=308)
Diarrhoea (Gastrointestinal disorders) | 17 (22) | 24 (26)
Hypertension (Vascular disorders) | 14 (14) | 21 (27)
Oedema peripheral (General disorders) | 21 (23) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03409107/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03409107/SAP_001.pdf